CLINICAL TRIAL: NCT06209801
Title: Comparison of the Effects of Mirror Therapy Integrated with Electrical Stimulation and Motor Imagery on Cortical Modulations in Patients with Peripheral Nerve Injury and Healthy Adults
Brief Title: Mirror Therapy Integrated with Electrical Stimulation for Cortical Modulations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202301500A3
Record Dates: First submitted 2024-01-03; First posted 2024-01-18 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Nerve Injuries
Keywords: mirror therapy; electrical stimulation; cortical modulation; motor imagery
MeSH Terms: conditions — Peripheral Nerve Injuries | interventions — Mirror Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Individuals with peripheral nerve injuries
  Interventions: Behavioral: Mirror therapy; Device: Neuromuscular electrical stimulation; Behavioral: Motor imagery
- Control group (Active Comparator): Healthy individuals
  Interventions: Behavioral: Mirror therapy; Device: Neuromuscular electrical stimulation; Behavioral: Motor imagery

INTERVENTIONS:
Behavioral: Mirror therapy — 60 seconds of intervention
Device: Neuromuscular electrical stimulation — 60 seconds of intervention
Behavioral: Motor imagery — 60 seconds of intervention

SUMMARY:
Peripheral nerve injury is common and can result in loss of sensation and motor function, reduced quality of life, and prolonged time to return to work. Maladaptive cortical reorganization occurs after nerve injury or immobilization and can further impair the recovery process. To improve the sensorimotor prognosis of people with peripheral nerve injury, methods such as mirror therapy, motor imagery, and electrical stimulation have been used in addition to usual care. However, no studies have shown the effect of integrating mirror therapy, motor imagery, and electrical stimulation in these individuals. Furthermore, the real-time effect of mirror therapy on cortical activation in this population remains unexplored. This study aims to determine the real-time cortical modulation effects of mirror therapy combined with electrical stimulation in individuals with peripheral nerve injury.

DETAILED DESCRIPTION:
Two groups of subjects (a group of peripheral nerve injury group and a group of healthy adults) will perform hand exercises in three randomized conditions: (1) mirror therapy with electrical stimulation and motor imagery, (2) electrical stimulation and motor imagery, and (3) motor imagery. Each participant performs specific sets of two exercises based on the type of nerve injury: (1) Median nerve injury: Picking up and putting down a pen using the thumb and index finger, and picking up and putting down a marble using the thumb and little finger. (2) Ulnar nerve injury: Picking up and putting down a card using the thumb and index finger, and picking up and putting down a marble using the thumb and little finger.(3) Brachial plexus injury: Picking up and putting down an empty cup, and picking up and putting down a pair of pliers. For combined median nerve and ulnar nerve injuries and healthy adult groups, movements corresponding to median nerve injuries are performed. Each experimental condition consists of 20 repetitions, lasting 60 seconds, followed by a 30-second rest between conditions. Relative alpha and beta band power in the sensorimotor cortex will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed median or ulnar nerve transection injury of the forearm in the past 6 months
* sufficient communication in the Chinese language
* being able to follow instructions
* muscle atrophy or lack of voluntary contraction over the injured hand, with maximum voluntary isometric contraction (MVIC) recorded with surface electromyography (EMG) less than 10% compared to the non-affected hand
* achieve an average score of 2 or above in the Kinesthetic and Visual Imagery Questionnaire-10 (KVIQ-10) for kinesthetic imagery

Exclusion Criteria:

* had central nervous disease
* had a recent (1 year) history of nerve entrapment syndrome
* had a history of latent neuropathy, such as diabetes or dialysis

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-11-21 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Relative alpha-band power in sensorimotor cortex | 10 minutes after the intervention
  Expressed as a percentage
Relative beta-band power in sensorimotor cortex | 10 minutes after the intervention
  Expressed as a percentage

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Hsia Chen, PhD, Principal Investigator — National Taiwan University, School of Medicine
Locations (2):
- Taiwan (2):
  - National Taiwain Univeristy, Colledge of Medicine, School and Graduate Institude of Physicl Therapy, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rizzo M, Petrini L, Del Percio C, Lopez S, Arendt-Nielsen L, Babiloni C. Mirror visual feedback during unilateral finger movements is related to the desynchronization of cortical electroencephalographic somatomotor alpha rhythms. Psychophysiology. 2022 Dec;59(12):e14116. doi: 10.1111/psyp.14116. Epub 2022 Jun 3. PMID 35657095
- [Background] Bello UM, Kranz GS, Winser SJ, Chan CCH. Neural Processes Underlying Mirror-Induced Visual Illusion: An Activation Likelihood Estimation Meta-Analysis. Front Hum Neurosci. 2020 Jul 31;14:276. doi: 10.3389/fnhum.2020.00276. eCollection 2020. PMID 32848663
- [Background] Binder E, Dovern A, Hesse MD, Ebke M, Karbe H, Saliger J, Fink GR, Weiss PH. Lesion evidence for a human mirror neuron system. Cortex. 2017 May;90:125-137. doi: 10.1016/j.cortex.2017.02.008. Epub 2017 Feb 24. PMID 28391066
- [Background] Cengiz B, Vuralli D, Zinnuroglu M, Bayer G, Golmohammadzadeh H, Gunendi Z, Turgut AE, Irfanoglu B, Arikan KB. Analysis of mirror neuron system activation during action observation alone and action observation with motor imagery tasks. Exp Brain Res. 2018 Feb;236(2):497-503. doi: 10.1007/s00221-017-5147-5. Epub 2017 Dec 11. PMID 29230518
- [Background] Scott M, Taylor S, Chesterton P, Vogt S, Eaves DL. Motor imagery during action observation increases eccentric hamstring force: an acute non-physical intervention. Disabil Rehabil. 2018 Jun;40(12):1443-1451. doi: 10.1080/09638288.2017.1300333. Epub 2017 Mar 21. PMID 28322596
- [Background] Zhang JJQ, Fong KNK, Welage N, Liu KPY. The Activation of the Mirror Neuron System during Action Observation and Action Execution with Mirror Visual Feedback in Stroke: A Systematic Review. Neural Plast. 2018 Apr 24;2018:2321045. doi: 10.1155/2018/2321045. eCollection 2018. PMID 29853839
- [Background] Bello UM, Winser SJ, Chan CCH. Role of kinaesthetic motor imagery in mirror-induced visual illusion as intervention in post-stroke rehabilitation. Rev Neurosci. 2020 Aug 27;31(6):659-674. doi: 10.1515/revneuro-2019-0106. PMID 32229682
- [Background] Wang J, Fritzsch C, Bernarding J, Holtze S, Mauritz KH, Brunetti M, Dohle C. A comparison of neural mechanisms in mirror therapy and movement observation therapy. J Rehabil Med. 2013 Apr;45(4):410-3. doi: 10.2340/16501977-1127. PMID 23474778
- [Background] Yang YJ, Jeon EJ, Kim JS, Chung CK. Characterization of kinesthetic motor imagery compared with visual motor imageries. Sci Rep. 2021 Feb 12;11(1):3751. doi: 10.1038/s41598-021-82241-0. PMID 33580093
- [Background] Chen YH, Siow TY, Wang JY, Lin SY, Chao YH. Greater Cortical Activation and Motor Recovery Following Mirror Therapy Immediately after Peripheral Nerve Repair of the Forearm. Neuroscience. 2022 Jan 15;481:123-133. doi: 10.1016/j.neuroscience.2021.11.048. Epub 2021 Dec 5. PMID 34875363
- [Background] Lu Y, Liu H, Hua X, Xu JG, Gu YD, Shen Y. Attenuation of brain grey matter volume in brachial plexus injury patients. Neurol Sci. 2016 Jan;37(1):51-56. doi: 10.1007/s10072-015-2356-1. Epub 2015 Aug 9. PMID 26255300
- [Background] Saavedra-Garcia A, Moral-Munoz JA, Lucena-Anton D. Mirror therapy simultaneously combined with electrical stimulation for upper limb motor function recovery after stroke: a systematic review and meta-analysis of randomized controlled trials. Clin Rehabil. 2021 Jan;35(1):39-50. doi: 10.1177/0269215520951935. Epub 2020 Aug 24. PMID 32830512